CLINICAL TRIAL: NCT04114669
Title: Behavioral Economics Trial To Enhance Regulation of Blood Pressure
Brief Title: Behavioral Economics Trial To Enhance Regulation of Blood Pressure (BETTER-BP)
Acronym: BETTER-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00952
Record Dates: First submitted 2019-09-20; First posted 2019-10-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regret lottery (Experimental): Will receive a lottery incentive ("regret lottery") for 6 months
  Interventions: Behavioral: Regret Lottery
- Control Condition (Placebo Comparator): Will complete a total of 3 in-person study visits, approximately one hour each.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Control Condition — 3 in-person study visits, approximately one hour each. These will take place at baseline, 6 months, and 12 months.
  Arms: Control Condition
Behavioral: Regret Lottery — Delivered by the Way to Health platform, installed on a smartphone and communicates with participants via text message.Participants are eligible to receive a potential cash reward if they are adherent with their antihypertensive medication the day before, which is monitored via electronic monitoring device (EMD) from AdhereTech. Each participant is assigned a 2-digit number for the trial, and each day the Way to Health platform randomly generates a 2-digit number. Participants will receive a prize if both digits match (1 in 100 chance) and will receive a prize of lesser value if one digit matches (18 in 100 chance). If they are not adherent with their medication, but would have won if they were adherent, they receive a text message that they would have won ("regret" component).
  Arms: Regret lottery

SUMMARY:
BETTER-BP (Behavioral Economics Trial To Enhance Regulation of Blood Pressure) is a phase II, single-center, prospective, pragmatic randomized clinical trial within the New York City Health and Hospitals (NYC-H+H) system and NYU Langone Family Health Centers. The trial will recruit from 3 NYC-H+H ambulatory clinics as well as NYU Langone Family Health Centers, and will use a lottery incentive program to promote adherence to antihypertensive medication that will be delivered via smartphone for 6 months. The trial will randomize 435 patients with hypertension determined to have poor adherence (<80% adherence with antihypertensive medication), in a 2:1 (intervention:control) ratio. Baseline enrollment will occur over 36 months with an expected 12 months follow-up per participant.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of hypertension.
* An active prescription for ≥1 antihypertensive medication (any of the following classes: thiazide diuretic, ACE inhibitor, angiotensin receptor blocker, beta blocker, calcium channel blocker, centrally acting alpha agonist, direct vasodilator).

  * 1 ambulatory systolic blood pressure ≥140 mmHg (on therapy).
* Suboptimal adherence (self-report).

Exclusion Criteria:

* Incarcerated
* Pregnant
* Unable to use study software (Way To Health) in English or Spanish
* Unable/unwilling to consent
* Clear barrier to technology use (e.g. visual or hearing impairment)
* Projected life expectancy <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) | Baseline, Month 6
  Three seated BPs will be measured after a rest period (5 minutes) using an automated device (Omron, Lake Forest, IL) which will reduce the potential for observer bias.

SECONDARY OUTCOMES:
Antihypertensive Adherence | Baseline, Month 6
  Measured with a wireless Tech wireless which transfers data via cell phone to the Way to Health platform. Adherence is measured as percentage of participants who "adhere" to treatment plan, defined as ≥ 80% of days covered.

CONTACTS AND LOCATIONS:
Overall Officials: John Dodson, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT04114669/ICF_000.pdf